CLINICAL TRIAL: NCT06771388
Title: Efficacy Evaluation of Avance QQ Collagen for Skin Beautification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-088-B
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Skin Condition; Liposomal Encapsulation
Keywords: Avance QQ Collagen; Double Nutri
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Non-liposomal collagen drink (Active Comparator)
  Interventions: Dietary Supplement: Non-liposomal collagen drink
- Liposomal collagen drink (Experimental)
  Interventions: Dietary Supplement: Liposomal collagen drink

INTERVENTIONS:
Dietary Supplement: Liposomal collagen drink — consume 50 g liquid drink daily for 8 consecutive weeks
  Other Names: Avance QQ Collagen
  Arms: Liposomal collagen drink
Dietary Supplement: Non-liposomal collagen drink — consume 50 g liquid drink daily for 8 consecutive weeks
  Arms: Non-liposomal collagen drink
Dietary Supplement: Placebo drink — consume 50 g liquid drink daily for 8 consecutive weeks
  Arms: Placebo drink

SUMMARY:
To assess Avance QQ Collagen product on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, age above 18 years old;
* The grade of crow's feet above 2 (Han et al. Sci Rep 13, 18903 (2023));
* Commitment not to use products having activity comparable with that of the product to be tested during the study period;
* Free of any dermatological or systemic disorder that would interfere with results.

Exclusion Criteria:

* Subject with obvious skin surface damage;
* Subject who had oral or topical medication which may affect skin condition within 1 month;
* Subject who is a vegetarian or likely to be acutely allergic to the listed ingredients in the product;
* Female who is pregnant, nursing or planning to become pregnant during the course of the study;
* Received facial laser therapy, chemical peeling in the past 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin collagen density. Units: arbitrary units
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  VISIA Complexion Analysis was utilized to measure skin wrinkles. Units: the amount of detectable wrinkles
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Cutometer® MPA580 was utilized to measure skin elasticity. Units: arbitrary units

SECONDARY OUTCOMES:
The change of wrinkles around the eyes | Change from Baseline wrinkles around the eyes at 8 weeks
  VISIA Complexion Analysis was utilized to measure wrinkles around the eyes. Units: the amount of detectable wrinkles
The change of skin hydration | Change from Baseline skin hydration at 8 weeks
  Corneometer® CM825 (CK, Germany) was utilized to measure skin surface hydation. Units: arbitrary Corneometer® units 0-120.
The change of skin lightness | Change from Baseline skin lightness at 8 weeks
  Chroma Meter MM500 was utilized to measure face skin lightness. Units: L* index
The change of skin tone | Change from Baseline skin tone at 8 weeks
  Chroma Meter MM500 was utilized to measure face skin color. Units: Individual Typology Angle (ITA°)

OTHER OUTCOMES:
The change of self-assessment skin condition | Change from Baseline skin condition at 8 weeks
  A self-assessment questionnaire was collected and evaluate skin condition.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Ph.D., Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Pingtung City, Taiwan